CLINICAL TRIAL: NCT04327505
Title: A Randomized, Controlled, Open Label, Multicentre Clinical Trial to Explore Safety and Efficacy of Hyperbaric Oxygen for Preventing ICU Admission, Morbidity and Mortality in Adult Patients With COVID-19
Brief Title: Safety and Efficacy of Hyperbaric Oxygen for ARDS in Patients With COVID-19
Acronym: COVID-19-HBO
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Futility, change of disease due to virus mutations and/or vaccination
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska Trial Alliance (Industry); University of California, San Diego (Other); Blekinge County Council Hospital (Other); JK Biostatistics AB (Unknown); The Swedish Research Council (Other Government); University of Regensburg (Other)
Responsible Party: Principal Investigator, Anders Kjellberg, MD, ICU Consultant/PhD student, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVID-19-HBO; 2020-001349-37 (EudraCT Number); K-1199/2020 (Registry Identifier: Karolinska Institutet)
Record Dates: First submitted 2020-03-25; First posted 2020-03-31 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: SARS (Severe Acute Respiratory Syndrome); Cytokine Storm; ARDS, Human; COVID-19; Sars-CoV2; Acute Respiratory Failure
Keywords: COVID-19; Hyperbaric oxygen; ARDS; SARS-CoV-2; ICU admission
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Cytokine Release Syndrome; Respiratory Distress Syndrome; COVID-19 | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: Randomized controlled, open label, multi-centre clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperbaric oxygen (Experimental): Hyperbaric oxygen 1,6-2.4 Bar for 30-60 minutes (compression/decompression time, according to local routines) in addition to best practice
  Interventions: Drug: Hyperbaric oxygen
- Control (No Intervention): Best practice

INTERVENTIONS:
Drug: Hyperbaric oxygen — 1.6- 2.4 ATA, 30-60 min (excluding compression/recompression)
  Other Names: HBO
  Arms: Hyperbaric oxygen

SUMMARY:
COVID-19 may cause severe pneumonitis that require ventilatory support in some patients, the ICU mortality is as high as 62%. Hospitals do not have enough ICU beds to handle the demand and to date there is no effective cure.

We explore a treatment administered in a randomized clinical trial that could prevent ICU admission and reduce mortality.

The overall hypothesis to be evaluated is that HBO reduce mortality, increase hypoxia tolerance and prevent organ failure in patients with COVID19 pneumonitis by attenuating the inflammatory response.

DETAILED DESCRIPTION:
Main objective: To evaluate if HBO reduce the number of ICU admissions compared to Best practice for COVID-19

Secondary objectives:

Main secondary objectives:

To evaluate if HBO:

* reduces mortality in severe cases of COVID-19.
* reduces morbidity associated with COVID-19.
* reduce the load on ICU resources in COVID-19.
* mitigate the inflammatory reaction in COVID-19.

Other secondary objectives (in selection):

To evaluate if HBO is safe for SARS-CoV-2 positive patients and staff.

Study design: Randomized, controlled, phase II, open label, multicentre

Study population: Adult patients with SARS-CoV-2 infection, with at least two risk factor for increased mortality, likely to develop ARDS criteria and need intubation within 7 days of admission to hospital.

Number of subjects: 200 (20+180)

Investigational product: Hyperbaric oxygen (HBO) compared with best practice treatment HBO: HBO 1.6-2.4 ATA for 30-60 min, maximum 5 treatments first 7 days Control: Best practice treatment for COVID-19

ELIGIBILITY:
Inclusion criteria:

1. Aged 18-90 years
2. PaO2/FiO2 (PFI) below 200 mmHg (26.7 kPa)
3. Suspected or verified SARS-CoV-2 infection
4. At least two risk factors for increased morbidity/mortality

   * Age above 50 years
   * Hypertension
   * Cardiovascular disease
   * Diabetes or pre-diabetes
   * Active or cured cancer
   * Asthma/COPD
   * Smoking
   * D-Dimer > 1.0 mg/L
   * Auto-immune disease
5. Documented informed consent according to ICH-GCP and national regulations

Exclusion Criteria:

1. ARDS/pneumonia caused by other viral infections (positive for other virus)
2. ARDS/pneumonia caused by other non-viral infections or trauma
3. Known pregnancy or positive pregnancy test in women of childbearing age
4. Patients with previous lung fibrosis more than 10%
5. CT- or Spirometry-verified severe COPD with Emphysema
6. Contraindication for HBO according to local guidelines
7. Not likely to need ICU admission < 7 days of screening (Subjective criteria that may exclude any patients that fulfil the other inclusion criteria but where the treating physician suspect a spontaneous recovery)
8. Mental inability, reluctance or language difficulties that result in difficulty understanding the meaning of study participation
9. Prisoner (Exclusion criteria according to IRB at UCSD)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adults, all genders
Enrollment: 34 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
ICU admission | Through study completion 30 days
  The proportion of subjects admitted to ICU from day 1 to day 30, based on at least one of the following criteria:
  i) Rapid progression over hours ii) Lack of improvement on high flow oxygen >40L/min or non invasive ventilation with fraction of inspired oxygen (FiO2) > 0.6 iii) Evolving Hypercapnia or increased work of breathing not responding to increased oxygen despite maximum standard of care available outside ICU iv) Hemodynamic instability or multi organ failure with maximum standard of care available outside ICU

SECONDARY OUTCOMES:
30-day mortality | Through study completion 30 days
  Proportion of subjects with 30-day mortality, all cause Mortality, from day 1 to day 30.
Time-to-intubation | Through study completion 30 days
  Time-to-Intubation, i.e. cumulative days free of invasive mechanical ventilation, from day 1 to day 30
Time-to-ICU | Through study completion 30 days
  Time-to-ICU, i.e. cumulative ICU free days, derived as the number of days from day 1 to ICU, where all ICU free subjects are censored at day 30.
Inflammatory response | Through study completion 30 days
  Mean change in inflammatory response from day 1 to day 30.
  1. White cell count + differentiation
  2. Procalcitonin
  3. C-Reactive protein
  4. Cytokines (IL-6) (if available at local laboratory)
  5. Ferritin
  6. D-Dimer
  7. LDH
Overall survival | Through study completion 30 days
  Overall survival (Kaplan-Meier)

OTHER OUTCOMES:
Hospital mortality | Through study completion 30 days
  Hospital mortality of any cause, proportion of subjects, from day 1 to day 30.
ICU mortality | From ICU admission to study completion 30 days
  Proportion of subjects with ICU mortality, Mortality of any cause in ICU, from day 1 to day 30.
Time in Invasive Ventilation | From ICU admission to study completion 30 days
  Time-to-stop of intubation/invasive mechanical ventilation, from ICU admission to day 30.
NEWS | Through study completion 30 days
  Mean daily NEWS from day 1 to day 30.
PaO2/FiO2 (PFI) | Through study completion 30 days
  Mean change in PaO2/FiO2 (PFI), from day 1 to day 2, … to day 30.
HBO Compliance | Day 1 to day 7
  1. Proportion of HBO treatments given vs planned.
  2. Proportion of subjects with HBO treatment administered within 24h after enrolment.
Hospital discharge | Through study completion 30 days
  Time-to-discharge from hospital
Oxygen dose | Through study completion 30 days
  Mean oxygen dose per day including HBO and cumulative pulmonary oxygen toxicity expressed as Units of oxygen pulmonary toxicity dose (UPTD) and Cumulative pulmonary toxicity dose (CPTD) from day 1 to day 30.
HBO dose | Day 1 to day 7
  Median number of HBO treatments and dose of HBO given, from day 1 to day 7
Micro RNA | Through study completion 30 days
  Change in expression of Micro RNA in plasma from day 1 to day 30
Hypoxic response | Through study completion 30 days
  Change in gene expression and Micro RNA interactions in Peripheral Blood Mononuclear Cells (PBMC) (20 Subjects) from day 1 to day 30
Immunological response | Through study completion 30 days
  Immunological response (20 subjects) from day 1 to day 30 in the following.
  1. Cytokines extended including (IL-1β, IL-2, IL-6, IL33 and TNFα)
  2. Lymphocyte profile
  3. Flowcytometry with identification of monocyte/lymphocyte subsets including but not limited to CD3+/CD4+/CD8+ and CD4+/CD8+ ratio
  4. FITMaN panel/Flow cytometry, Interleukins (IL-1β, IL-2, IL-6, IL33 and TNFα),
  5. T-reg cells (CD3+/CD4+/CD25+/CD127+)
  6. Monocyte proliferation markers, Ex vivo monocyte function
Multi organ dysfunction | Through study completion 30 days
  Mean change in routine biomarkers for organ dysfunction, from day 1to day 30.
Viral load | Through study completion 30 days
  Viral load, review of records from day 1 to day 30.
Secondary infections | Through study completion 30 days
  Number of secondary infections, review of records, number of events and patients from day 1 to day 30.
Pulmonary embolism | Through study completion 30 days
  Diagnosed PE needing treatment, review of records, number of events and patients from day 1 to day 30.
Pulmonary CT | Through study completion 30 days
  Changes on Pulmonary CT, review of records from day 1 to day 30.
Chest X-ray | Through study completion 30 days
  Changes on Chest X-ray, review of records from day 1 to day 30.
Lung ultrasound | Through study completion 30 days
  Changes in Lung ultrasound, review of records from day 1 to day 30.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Kjellberg, MD, Principal Investigator — Karolinska Institutet; Peter Lindholm, MD, PhD, Study Chair — Karolinska Institutet; Kenny Rodriguez-Wallberg, MD, PhD, Study Chair — Karolinska Institutet
Locations (3):
- Krankenhaus St. Joesf, Regensburg, Germany
- Sweden (2):
  - Blekingesjukhuset, Karlskrona, Blekinge County
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
The full study protocol, statistical plan and consent form will be publicly available when results are published. Data will be available on patient level; data will be pseudonymized. The full dataset and statistical code will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting after publication and for 36 months
Access Criteria: A full description of the intended use of the data must be sent to the corresponding author for review and approval. Participant consent for data sharing is conditioned and new ethics approval may be required.

REFERENCES:
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Oscarsson N, Muller B, Rosen A, Lodding P, Molne J, Giglio D, Hjelle KM, Vaagbo G, Hyldegaard O, Vangedal M, Salling L, Kjellberg A, Lind F, Ettala O, Arola O, Seeman-Lodding H. Radiation-induced cystitis treated with hyperbaric oxygen therapy (RICH-ART): a randomised, controlled, phase 2-3 trial. Lancet Oncol. 2019 Nov;20(11):1602-1614. doi: 10.1016/S1470-2045(19)30494-2. Epub 2019 Sep 16. PMID 31537473
- [Background] Thibodeaux K, Speyrer M, Raza A, Yaakov R, Serena TE. Hyperbaric oxygen therapy in preventing mechanical ventilation in COVID-19 patients: a retrospective case series. J Wound Care. 2020 May 1;29(Sup5a):S4-S8. doi: 10.12968/jowc.2020.29.Sup5a.S4. PMID 32412891
- [Background] Gorenstein SA, Castellano ML, Slone ES, Gillette B, Liu H, Alsamarraie C, Jacobson AM, Wall SP, Adhikari S, Swartz JL, McMullen JJS, Osorio M, Koziatek CA, Lee DC. Hyperbaric oxygen therapy for COVID-19 patients with respiratory distress: treated cases versus propensity-matched controls. Undersea Hyperb Med. 2020 Third Quarter;47(3):405-413. doi: 10.22462/01.03.2020.1. PMID 32931666
- [Background] Kjellberg A, De Maio A, Lindholm P. Can hyperbaric oxygen safely serve as an anti-inflammatory treatment for COVID-19? Med Hypotheses. 2020 Nov;144:110224. doi: 10.1016/j.mehy.2020.110224. Epub 2020 Aug 30. PMID 33254531
- [Derived] Kjellberg A, Douglas J, Hassler A, Al-Ezerjawi S, Bostrom E, Abdel-Halim L, Liwenborg L, Hetting E, Jonasdottir Njastad AD, Kowalski J, Catrina SB, Rodriguez-Wallberg KA, Lindholm P. COVID-19-Induced Acute Respiratory Distress Syndrome Treated with Hyperbaric Oxygen: Interim Safety Report from a Randomized Clinical Trial (COVID-19-HBO). J Clin Med. 2023 Jul 24;12(14):4850. doi: 10.3390/jcm12144850. PMID 37510965
- [Derived] Kjellberg A, Douglas J, Pawlik MT, Kraus M, Oscarsson N, Zheng X, Bergman P, Franberg O, Kowalski JH, Nyren SP, Silvanius M, Skold M, Catrina SB, Rodriguez-Wallberg KA, Lindholm P. Randomised, controlled, open label, multicentre clinical trial to explore safety and efficacy of hyperbaric oxygen for preventing ICU admission, morbidity and mortality in adult patients with COVID-19. BMJ Open. 2021 Jul 5;11(7):e046738. doi: 10.1136/bmjopen-2020-046738. PMID 34226219
- See also: Hyperbaric medicine research group, Karolinska Institutet — https://ki.se/en/fyfa/hyperbaric-medicine
- See also: COVID-19 EUBS-ECHM position statement on HBOT — http://www.eubs.org/?p=1074
- See also: KI News-description of trial in layman language — https://news.ki.se/ki-researchers-to-evaluate-effect-of-hyperbaric-oxygen-treatment-against-covid-19